CLINICAL TRIAL: NCT06282991
Title: Lorlatinib in Patients With Advanced Non-Small Cell Lung Cancer Who Progress on First- and Second- Generation Tyrosine Kinase Inhibitor: A Real-world Evidence Among Taiwanese Population, Non-Interventional Study
Brief Title: A Study to Learn About Lorlatinib in Patients With Non-Small Cell Lung Cancer Which Could Not Be Controlled
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B7461028
Record Dates: First submitted 2024-02-01; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Non-Small Cell Lung Carcinoma
Keywords: ALK; TKI; Lorlatinib; RWE
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — lorlatinib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lorlatinib: Patients received lorlatinib treatment under EAP
  Interventions: Drug: Lorlatinib

INTERVENTIONS:
Drug: Lorlatinib — ALK/ROS1 tyrosine kinase inhibitor
  Other Names: PF-6463992

SUMMARY:
The purpose of this study is to learn about lorlatinib for the possible treatment of lung cancer which could not be controlled.

This study is seeking participants who:

* have lung cancer that could not be controlled.
* have a type of gene called anaplastic lymphoma kinase. A gene is a part of your DNA that has instructions for making things your body needs to work.
* have received at least 1 treatment before.

All participants in this study had received lorlatinib. Lorlatinib is a tablet that is taken by mouth at home. They continued to take dacomitinib until their cancer was no longer responding. The study will look at the experiences of people receiving the study medicine. This will help to see if the study medicine is safe and effective.

DETAILED DESCRIPTION:
Non-small cell lung cancer (NSCLC; 80-85% of all lung cancers) remains the most common cause of cancer-related mortality globally, most often diagnosed in advanced stages. Targeted drugs are currently the most often used therapies for advanced NSCLC patients that harbor molecular alterations, including the echinoderm microtubule-associated protein like 4 (EML4)-anaplastic lymphoma kinase (ALK) translocation. For ALK-positive NSCLC patients, crizotinib, ceritinib, alectinib, and brigatinib, are the first- and second-generation tyrosine kinase inhibitors (TKIs). Although the benefit of them has been demonstrated in series of pivotal clinical trials, most patients who initially derive the benefit latterly develop resistance due to secondary mutations. Lorlatinib, a third-generation inhibitor, is a TKI of ALK and Receptor Tyrosine Kinase C-Ros Oncogene I (ROS-1). It is also a potent TKI that is effectively against known resistant mutants that mediate resistance to first- and second-generation ALK-TKIs. Despite the efficacy and safety data derived from the pivotal phase I/II clinical trial, there are limited data describing the use of lorlatinib and its outcomes in real-world practice settings outside the highly controlled environs of clinical trials. The objective of this study is therefore to evaluate real-world systemic treatment patterns, clinical outcome, therapeutic effect, safety profile of Lorlatinib in advanced NSCLC patients, and also factors associated with clinical outcome in those Lorlatinib treated patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years old
* Patients who were approved to join Lorlatinib CUP on or before 31 Jul 2019 while initiate Lorlatinib treatment before 30 Sep 2019,
* Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Patient treated Lorlatinib other than CUP.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects will be enrolled from Lorlatinib Compassionate Use Program (CUP) and should be entered into this observational study at the physician's discretion.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2021-01-18 (Actual); Study Completion 2021-01-18 (Actual)

PRIMARY OUTCOMES:
The treatment pattern from initial diagnosis to current lorlatinib treatment. | 1 year prior to lorlatinib treatment started
  To describe the treatment from initial diagnosis of NSCLC and the line setting of lorlatinib for their metastatic NSCLC with ALK or ROS1 rearrangement

SECONDARY OUTCOMES:
objective response rate (ORR) | From first dose of lorlatinib until 30 Sep 2020 or death whichever occurred first, assessed upto 30 months.
  Percentage of the best response recorded for each participants during lorlatinib treatment.
overall survival | From first dose of lorlatinib until 30 Sep 2020 or death whichever occurred first, assessed upto 30 months.
  duration (month) between first dose of lorlatinib and death or end of study
progression-free survival | From first dose of lorlatinib until 30 Sep 2020, or first documented progression or date of death from any cause, whichever came first, assessed upto 30 months.
  duration (month) between first dose of lorlatinib and disease progression or death or end of study
1-year OS rate | from first dose of lorlatinib to 12 months later
  percentage of survival in first year
time-to-treatment failure for all NSCLC | From first dose of lorlatinib until 30 Sep 2020 or death from any cause, whichever occurred first, assessed up to 30 months.
  duration of treatment of all NSCLC treatment captured from medical records
time-to-treatment failure of lorlatinib | From first dose of lorlatinib until 30 Sep 2020 or death whichever occurred first, assessed upto 30 months.
  duration (month) between lorlatinib start and disease progression by investigator's final assessment
The clinical nature, incidence, duration, and severity of lorlatinib-related safety profile | From first dose of lorlatinib until 30 Sep 2020 or death whichever occurred first, assessed upto 30 months.
  The clinical nature, incidence, duration, and severity of Lorlatinib related adverse drug reaction; outcome and possible causality will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- Taiwan (6):
  - CHANG GUNG MEMORIAL HOSPITAL Kaohsiung Branch, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital - Linkou Branch, Taoyuan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7461028